CLINICAL TRIAL: NCT01699061
Title: A PHASE 1 SINGLE-BLIND, SINGLE-SEQUENCE STUDY ASSESSING THE EFFECT OF TIVANTINIB ON THE QTC INTERVAL IN CANCER SUBJECTS
Brief Title: Effect of Tivantinib on the QTC Interval in Cancer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ARQ197-A-U159
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2018-02

CONDITIONS: Solid Tumors
MeSH Terms: interventions — ARQ 197

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablet administered with a meal twice a day on Day 1
  Interventions: Drug: Placebo
- Tivantinib (Experimental): 3 tivantinib tablets 120 mg administered twice daily with a meal starting on Day 2
  Interventions: Drug: Tivantinib

INTERVENTIONS:
Drug: Tivantinib — 3 tivantinib tablets 120 mg administered twice daily with a meal starting on Day 2
  Other Names: ARQ 197
  Arms: Tivantinib
Drug: Placebo — Placebo tablet administered with a meal twice a day on Day 1
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of tivantinib on the QTc interval in patients with solid tumors

DETAILED DESCRIPTION:
The study is designed to estimate the maximum change in QTcF (change from baseline) between placebo and multiple-dose tivantinib. A tivantinib oral dose of 360 mg BID has been selected for this study because this is the highest dose currently being evaluated in clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a histologically or cytologically confirmed advanced solid tumor at Screening
* Male or female greater than or equal to 18 years of age
* Women of childbearing potential must have a negative pregnancy test performed prior to the start of study drug
* Subjects (male and female) of childbearing potential must agree to use double barrier contraceptive measures or avoid intercourse during the study and for 90 days after the last dose of study drug. In addition, all female subjects of childbearing potential must have a negative pregnancy test result before initiating study treatment
* An Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
* Adequate bone marrow and liver function, defined as:
* Platelet count greater than or equal to 100 × 109/L
* Hemoglobin greater than or equal to 9.0 g/dL
* Absolute neutrophil count greater than or equal to 1.5 × 109/L
* Total bilirubin less than or equal to 1.5 × upper limit of normal (ULN)
* Alanine aminotransferase and aspartate aminotransferase less than or equal to 3 × ULN (less than or equal to 5 × ULN for subjects with liver metastases)
* Serum creatinine less than or equal to 1.5 × ULN
* Electrolytes within normal limits, particularly potassium, magnesium, & calcium. Supplementation is permitted as needed
* Subjects should be able to provide written informed consent, comply with protocol visits and procedures, be able to take oral medication, and not have any active infection or chronic co-morbidity that would interfere with therapy
* Subjects must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an IRB-approved ICF (including HIPAA authorization, if applicable) before performance of any study-specific procedures or tests

Exclusion Criteria:

* History of cardiac disease:
* Active coronary artery disease, defined as myocardial infarction, unstable angina, coronary bypass graft, or stenting within 6 months prior to study entry
* Evidence of uncontrolled bradycardia or other cardiac arrhythmia defined as greater than or equal to Grade 2 according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4, or uncontrolled hypertension
* Any of the following ECG findings: PR interval greater than 240 msec or less than or equal to 110 msec or bradycardia defined as sinus rate <50 beats per minute
* Mean QTcF interval greater than 450 msec on triplicate centrally read Screening ECGs
* Cardiac conduction abnormalities denoted by any of the following: evidence of second-degree (type II) or third-degree atrioventricular block, evidence of ventricular pre-excitation, ECG evidence of complete left bundle branch block, intraventricular conduction delay with QRS duration greater than 120 msec, atrial fibrillation, or presence of cardiac pacemaker
* Personal or family history of long-QT syndrome
* Active, clinically serious infections defined as greater than or equal to Grade 2 according to NCI CTCAE, version 4
* Known metastatic brain or meningeal tumors, unless that subject is greater than 3 months from definitive therapy and clinically stable (supportive therapy with steroids or anticonvulsant medications is allowed) with respect to the tumor at the time of first dose of study drug
* Pregnant or breastfeeding
* Any major surgical procedure within 3 weeks prior to the first dose of study drug
* Significant gastrointestinal disorders, in the opinion of the Principal Investigator (eg, Crohn's disease, ulcerative colitis, extensive gastric resection, comorbid disease which causes malabsorption of the drug)
* Received tivantinib as prior therapy
* Received anticancer therapy, including antibody, retinoid, or hormonal treatment (except megestrol acetate as supportive care), and radiation, within 3 weeks before dosing. Prior and concurrent use of hormone replacement therapy, the use of gonadotropin-releasing hormone modulators for prostate cancer, and the use of somatostatin and analogs for neuroendocrine tumors are permitted
* Any other investigational drug within 3 weeks prior to dosing
* Substance abuse or medical, psychological, or social conditions that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results
* Any condition that is unstable or that could jeopardize the safety of the subject and the subject's protocol compliance, including known infection with human immunodeficiency virus, hepatitis B virus, or hepatitis C virus
* Inability to swallow oral medications that could interfere with the absorption of tivantinib
* Administration or possibility of initiating or continuing any treatment with any known CYP 3A4 and CYP2C19 enzyme and P-glycoprotein altering drugs (inducer or inhibitor) or non-drug agents or gastric pH modifiers within the 14 days prior to dosing and/or during the PK evaluation (14 to 15 days) after initiation of the study treatment
* Subjects with a clinical diagnosis of hepatic impairment and/or hepatocellular carcinoma and/or chronic liver cirrhosis with confirmation either by previous biopsy or with findings on ultrasound, computed tomography (CT) or MRI consistent with chronic liver cirrhosis
* Subjects who are on treatment receiving drugs that may affect QTc (eg, quinidine or moxifloxacin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2012-07; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The time-matched difference in the QTcF interval at each timepoint after both single and multiple doses of tivantinib compared with placebo | Baseline and 1, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 2, and 5 (+3 days)
  Triplicate ECG measurements of the QTc interval will be taken at Screening (4 sets each 1 hour apart) and pre-dose and 1, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 2, and 5 (+3 days)

SECONDARY OUTCOMES:
Estimated change in baseline adjusted QT, corrected QT interval (QTcB), individually corrected QT interval (QTcI) (if possible), heart rate, PR, QRS, & RR intervals at timepoints after both single and multiple doses of tivantinib compared with placebo | Baseline and 1, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 2, and 5 (+3 days)
  Triplicate ECG measurements of the QTc interval will be taken at Screening (4 sets each 1 hour apart) and pre-dose and 1, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 2, and 5 (+3 days)
Plasma pharmacokinetic (PK) profiles of tivantinib and major metabolites of tivantinib after both single and multiple doses of tivantinib. | Baseline and 1, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 2, and 5 (+3 days)
  Blood samples for PK analysis will be obtained within 15 minutes following each pre-specified ECG measurement
Explore the tivantinib plasma concentration-QTc interval relationship | Baseline and 1, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 2, and 5 (+3 days)
  Triplicate ECG measurements of the QTc interval will be taken at Screening (4 sets each 1 hour apart) and pre-dose and 1, 2, 3, 4, 6, 8, and 12 hours post dose on Days 1, 2, and 5 (+3 days). Blood samples for PK analysis will be obtained within 15 minutes following each pre-specified ECG measurement. The relationship between plasma concentrations of tivantinib and the change from baseline in QTc will be quantified using a linear random coefficient regression model approach.

CONTACTS AND LOCATIONS:
Overall Officials: Hamim Zahir, BPharm, PhD, Study Director — Daiichi Sankyo UK Ltd.
Locations (1):
- START - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/